CLINICAL TRIAL: NCT02116452
Title: Effects of GOS/PDX Supplemented Formula in Preventing and Modifying the History of Allergy and Acute Infections in a Population of Infants at Risk of Atopy
Brief Title: Prebiotics in Prevention of Atopy
Acronym: PIPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Alfredo Guarino, Head physician of Department of Translational Medical Science, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PIPA
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2011-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breast Milk (No Intervention): Breast FED newborns
- Standard Formula (Placebo Comparator): Standard Formula FED newborns
- Supplemented Formula (Active Comparator): GOS/PDX Formula FED newborns
  Interventions: Dietary Supplement: Supplemented Formula

INTERVENTIONS:
Dietary Supplement: Supplemented Formula — 50:50 mixture of GOS/PDX formula will be administered
  Arms: Supplemented Formula

SUMMARY:
The study objective is to evaluate whether a specific prebiotic (GOS/PDX) may have an effect in preventing atopic dermatitis, food allergy, intestinal and/or respiratory infections in infants at risk of atopy. In infants with dermatitis, the hypothesis will be tested that prebiotics reduce the severity of the disease.

DETAILED DESCRIPTION:
This study is a prospective, double blind, randomised, 24 month study trial comparing formula with 50/50 mixture of GOS/PDX (Enfamil Premium Infant Formula 1 for children <6 months and Formula 2 for children ≥ 6 months) versus standard formula (Enfamil Premium Formula 1 and 2).

Study population is composed by newborns at risk for allergy that will be identified at time of delivery. Infants will be eligible if at least one parent or one older sibling have a physician-diagnosed atopic disease (asthma, allergic rhinoconjunctivitis , atopic dermatitis, allergic urticaria, and food allergy as follow described. At time of enrolment (within the first 4 weeks of life) infants will be randomised 1:1 to receive once they will start formula feeding before the day of the 6th month birthday.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age >37 and < 42 weeks.
2. Birth weight > 2500 gr.
3. At risk of atopy (see appendix 1).
4. Informed consent signed by the parents (see appendix 3).

Exclusion Criteria:

1. Congenital immunodeficiency
2. Severe congenital disorders or malformations
3. Born to mother with diabet
4. Long term intake (> 7 consecutive days) of pro- or prebiotics
5. Children who have already assumed ≥ 50 mL for feeding bottle of Formulas different from the one object of this study for up to a month.
6. Parents expected not to be compliant with the study procedures

Ages: 1 Week to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence | 36 - 48 weeks
  Cumulative incidence of atopic dermatitis at 36 and 48 weeks

SECONDARY OUTCOMES:
Severity | 36-48 weeks
  Severity of atopic dermatitis as judged by the SCORAD score at 36 and 48 weeks and its distribution in three different groups: mild (<15 SCORAD points), moderate (15-40 SCORAD points), and severe (>40 SCORAD points) according to the objective components of the index

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Guarino, MD, Principal Investigator — University of Naples; Stefania Zanconato, MD, Principal Investigator — University of Padova
Locations (1):
- University of Padova - Department of Pediatrics, Padua, Italy, Italy

REFERENCES:
- [Derived] Ranucci G, Buccigrossi V, Borgia E, Piacentini D, Visentin F, Cantarutti L, Baiardi P, Felisi M, Spagnuolo MI, Zanconato S, Baraldi E, Giaquinto C, Guarino A. Galacto-Oligosaccharide/Polidextrose Enriched Formula Protects against Respiratory Infections in Infants at High Risk of Atopy: A Randomized Clinical Trial. Nutrients. 2018 Mar 1;10(3):286. doi: 10.3390/nu10030286. PMID 29494489